CLINICAL TRIAL: NCT02895932
Title: Serotonin and Amyloidopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Roger L. Albin, Principal Investigator, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00094478
Record Dates: First submitted 2015-12-01; First posted 2016-09-12 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case (Experimental): Patients with diagnosed Parkinson's disease
  Interventions: Radiation: PET imaging
- Control (Experimental): Healthy adults
  Interventions: Radiation: PET imaging

INTERVENTIONS:
Radiation: PET imaging — Serotonin, Dopamine and Amyloid PET imaging

SUMMARY:
The purpose of this study is to determine if changes in brain serotonin affects the accumulation of amyloid in the brain. The investigators will use brain imaging methods to measure the amount of serotonin and amyloid in the brain of individuals with Parkinson's Disease (PD) and otherwise healthy older people. PD participants will undergo repeat brain imaging to assess amyloid accumulation two years after their first brain imaging session. All participants will undergo examinations to assess their motor function, and asked questions to assess their mood and thinking.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common problem of older people often causing significant problems with thinking and memory. Abnormal accumulation within in the brain of a protein called amyloid is felt to contribute to impaired thinking and memory in PD. Excessive accumulation of this protein is also involved in Alzheimer disease (AD) and may influence thinking and memory in otherwise healthy older people. Recent evidence suggests that changes in the amount of another brain chemical, serotonin, influences the amount of amyloid accumulating in the brains of people with PD and otherwise healthy older people. The purpose of this study is to determine if changes in brain serotonin affects the accumulation of amyloid in the brain. The investigators use brain imaging methods to measure the amount of serotonin and amyloid in the brain of individuals with PD and otherwise healthy older people. PD participants will undergo repeat brain imaging to assess amyloid accumulation 2 years after their first brain imaging session. All participants will undergo examinations to assess their motor function, and asked questions to assess their mood and thinking.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have been diagnosed with Parkinson disease age 45 years and older are eligible to participate in this study.
* Healthy older individuals (ages 60-80) without neurologic problems are eligible to participate.

Exclusion Criteria:

* Individuals using some drugs cannot participate. These include anti-depressant medications, buproprion, or St. John's Wort, as well as dopamine antagonist medications.
* Women of childbearing age may not participate.
* Individuals unable to have MRI scans because of a pacemaker or metal fragments may not participate.
* Individuals with a history of stroke may not participate. People with any contraindication of PET imaging such as previous participation in research procedures involving ionizing radiation may not be eligible to participate in this study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Regional brain beta amyloid levels and regional brain serotonin terminal density as measured by PET brain imaging. | 2 years
  The PET imaging measures of regional brain beta amyloid levels and regional serotonin terminal density will be compared across participants to determine if there is a relationship between the regional density of serotonin terminals and the accumulation of beta amyloid.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States